CLINICAL TRIAL: NCT00296036
Title: A Phase III Randomized, Placebo-controlled, Double-blind Trial to Determine the Effectiveness of a Urea/Lactic Acid-Based Topical Keratolytic Agent and Vitamin B-6 for Prevention of Capecitabine-Induced Hand and Foot Syndrome
Brief Title: Pyridoxine and Topical Urea/Lactic Acid-Based Cream in Preventing Hand-Foot Syndrome in Patients Receiving Capecitabine for Breast Cancer or Other Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N05C5; NCI-2009-00655 (Registry Identifier: CTRP (Clinical Trials Reporting System)); ROCHE-NCCTG-N05C5; CDR0000464246 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer; Drug/Agent Toxicity by Tissue/Organ; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: drug/agent toxicity by tissue/organ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm I (closed to accrual as of 10/24/2007) (Experimental): Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily and oral pyridoxine once daily on days 1-21.
  Interventions: Dietary Supplement: pyridoxine hydrochloride; Drug: urea/lactic acid-based topical cream
- Arm II (closed to accrual as of 10/24/2007) (Experimental): Patients receive topical urea/lactic acid-based cream as in arm I (closed to accrual as of 10/24/2007) and oral placebo once daily on days 1-21.
  Interventions: Drug: urea/lactic acid-based topical cream; Other: placebo
- Arm III (closed to accrual as of 10/24/2007) (Experimental): Patients receive placebo cream applied to palms and soles twice daily and pyridoxine as in arm I (closed to accrual as of 10/24/2007).
  Interventions: Dietary Supplement: pyridoxine hydrochloride; Other: placebo
- Arm IV (closed to accrual as of 10/24/2007) (Placebo Comparator): Patients receive placebo cream as in arm III and oral placebo as in arm II (closed to accrual as of 10/24/2007).
  Interventions: Other: placebo
- Arm V (Experimental): Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily on days 1-21.
  Interventions: Drug: urea/lactic acid-based topical cream
- Arm VI (Placebo Comparator): Patients receive placebo cream applied to palms and soles twice daily on days 1-21.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: pyridoxine hydrochloride — Given orally
  Arms: Arm I (closed to accrual as of 10/24/2007); Arm III (closed to accrual as of 10/24/2007)
Drug: urea/lactic acid-based topical cream — Applied topically
  Arms: Arm I (closed to accrual as of 10/24/2007); Arm II (closed to accrual as of 10/24/2007); Arm V
Other: placebo — Given orally or applied topically
  Arms: Arm II (closed to accrual as of 10/24/2007); Arm III (closed to accrual as of 10/24/2007); Arm IV (closed to accrual as of 10/24/2007); Arm VI

SUMMARY:
RATIONALE: Pyridoxine (vitamin B6) and topical urea/lactic acid-based cream may prevent or lessen hand-foot syndrome caused by chemotherapy. It is not yet known whether giving pyridoxine with or without topical urea/lactic acid-based cream is more effective than topical urea/lactic acid-based cream alone or a placebo in preventing hand-foot syndrome.

PURPOSE: This randomized phase III trial is studying pyridoxine and topical urea/lactic acid-based cream to see how well they work compared with giving pyridoxine together with a placebo, giving topical urea/lactic acid-based cream together with a placebo, or giving two placebos in preventing hand-foot syndrome in patients who are receiving capecitabine for breast cancer or other cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the prophylactic use of a topical urea/lactic acid cream can decrease the incidence/severity of capecitabine-caused palmar-plantar erythrodysesthesia in patients receiving capecitabine for breast and/or other cancer.
* Evaluate the potential toxicity of this cream.
* Determine whether the prophylactic use of vitamin B6 can decrease the incidence and/or severity of capecitabine-caused palmar-plantar erythrodysesthesia.
* Evaluate the potential toxicity of vitamin B6.
* Determine whether the prophylactic use of a topical urea/lactic acid cream in combination with vitamin B6 can decrease the incidence and/or severity of capecitabine caused palmar-plantar erythrodysesthesia.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to age (< 50 years old vs 50-60 years old vs > 60 years old), sex, capecitabine dose level (2000 mg/day vs 2500 mg/day), cancer type (breast vs other), and mode of therapy (adjuvant [including neo-adjuvant] therapy vs metastatic disease). Patients are randomized to 1 of 6 treatment arms (treatment arms I-IV closed to accrual as of 10/24/007).

* Arm I (closed to accrual as of 10/24/2007): Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily and oral pyridoxine once daily on days 1-21.
* Arm II (closed to accrual as of 10/24/2007): Patients receive topical urea/lactic acid-based cream as in arm I (closed to accrual as of 10/24/2007) and oral placebo once daily on days 1-21.
* Arm III (closed to accrual as of 10/24/2007): Patients receive placebo cream applied to palms and soles twice daily and pyridoxine as in arm I (closed to accrual as of 10/24/2007).
* Arm IV (closed to accrual as of 10/24/2007):Patients receive placebo cream as in arm III and oral placebo as in arm II (closed to accrual as of 10/24/2007).
* Arm V: Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily on days 1-21.
* Arm VI: Patients receive placebo cream applied to palms and soles twice daily on days 1-21.

In all arms, treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast and/or other cancer
* Undergoing first treatment with capecitabine as adjuvant (including neo-adjuvant) therapy OR for metastatic disease

  * Receiving a dose of capecitabine either 2,000 mg/day (1,000 mg twice daily) OR 2,500 mg/day for 14 days with 4 courses of therapy at 3 week (+/- 3 days) intervals
* Hormone-receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* No history of allergy to urea-containing cream
* No pre-existing neuropathy ≥ grade 2
* No other dermatologic condition, that, in the opinion of the physician, may affect the hands or feet or may complicate evaluation during study treatment

PRIOR CONCURRENT THERAPY:

* No other concurrent agents that function to prevent palmar-plantar erythrodysesthesia caused by capecitabine or topical agents in the hands or feet for other indications (e.g., dryness)
* No concurrent vitamin B6 > 50 mg/day
* No concurrent or planned use of over-the-counter products that contain urea or lactic acid, including any of the following:

  * Aqua Care®
  * Medicated Calamine^® lotion (0.3%)
  * Coppertone^® Waterproof Ultra Protection Sunblock
  * Dr. Scholl's^® Smooth Touch deep moisturizing cream
  * Depicure^® So Smooth Cream
  * Dove^® Moisturizing Cream Wash
  * Cetaphil^ ®Moisturizing Cream
  * Vaseline Intensive Care ^ ® lotion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2006-06; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (231):
- United States (231):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Wolf SL, Qin R, Menon SP, Rowland KM Jr, Thomas S, Delaune R, Christian D, Pajon ER Jr, Satele DV, Berenberg JL, Loprinzi CL; North Central Cancer Treatment Group Study N05C5. Placebo-controlled trial to determine the effectiveness of a urea/lactic acid-based topical keratolytic agent for prevention of capecitabine-induced hand-foot syndrome: North Central Cancer Treatment Group Study N05C5. J Clin Oncol. 2010 Dec 10;28(35):5182-7. doi: 10.1200/JCO.2010.31.1431. Epub 2010 Nov 8. PMID 21060036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial was originally designed as a two-by-two factorial trial to test if urea/lactic acid-based cream and/or oral pyridoxine (B6) could decrease capecitabine-caused HFS. After results from another study found B6 and capecitabine combination ineffective in preventing HFS, the study was amended to a two-arm, randomized clinical trial.
Groups:
- Arm I: (Urea/Lactic Acid +Vit B6): Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily and oral pyridoxine once daily on days 1-21.
- Arm II: (Urea/Lactic Acid + Placebo): Patients receive topical urea/lactic acid-based cream as in arm I (closed to accrual as of 10/24/2007) and oral placebo once daily on days 1-21.
- Arm III: (Placebo +Vit B6): Patients receive placebo cream applied to palms and soles twice daily and pyridoxine as in Arm I
- Arm IV: (Placebo + Placebo): Patients receive placebo cream and oral placebo.
- Arm V: Urea/Lactic Acid: Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily on days 1-21.
- Arm VI: (Placebo): Patients receive placebo cream applied to palms and soles twice daily on days 1-21.
Period: Overall Study
Arm/Group | Arm I: (Urea/Lactic Acid +Vit B6) | Arm II: (Urea/Lactic Acid + Placebo) | Arm III: (Placebo +Vit B6) | Arm IV: (Placebo + Placebo) | Arm V: Urea/Lactic Acid | Arm VI: (Placebo)
Started | 19 | 18 | 18 | 17 | 33 | 32
Completed | 18 | 18 | 16 | 16 | 31 | 28
Not Completed | 1 | 0 | 2 | 1 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Arms I (18), II (18), and IV (31) were combined and analyzed as patients treated with Urea/Lactic Acid Cream. Arms III (16), IV (16), and VI (28) were combined as patients treated with placebo in place of Urea/Lactic Acid Cream.
Groups:
- Urea/Lactic Acid Cream: Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily on days 1-21.
- Placebo Cream: Patients receive placebo cream applied to palms and soles twice daily on days 1-21.
- Total: Total of all reporting groups
Arm/Group | Urea/Lactic Acid Cream | Placebo Cream | Total
Number analyzed (Participants) | 67 | 60 | 127
Age, Customized [Number; unit: participants]
  <50 | 11 | 9 | 20
  50-60 | 19 | 17 | 36
  > 60 | 37 | 34 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 101
  Male | 15 | 11 | 26
Region of Enrollment [Number; unit: participants]
  United States | 67 | 60 | 127

OUTCOME MEASURES:

1. Primary Outcome: To Determine Whether the Prophylactic Use of a Topical Urea/Lactic Acid Cream Can Decrease the Incidence/Severity of Capecitabine-caused Palmar-plantar Erythrodysesthesia
Description: A patient self-reported hand-foot syndrome (HFSD), also known as palmar-plantar erythrodysesthesia, was completed daily while applying the cream. Patients rated skin severity symptoms individually in their hands and in their feet. Definitions of symptoms, which were based on Common Terminology Criteria for Adverse Events (CTCAE) v3.0, were provided to patients. The number of patients reporting moderate to severe symptoms in either hands or feet were tabulated and percentages are reported.
Time Frame: First 3 weeks of treatment
Population: Eight patients from the Urea/Lactic Acid group were not included in the primary analysis (1 did not fill out the diary, 1 refused treatment, 3 had adverse events before completing the diary, and 3 for other reasons). For the placebo arm, 11 were excluded (2 refused further treatment, 2 had adverse events, and 7 went off for other reasons).
Measure: Number; unit: percentage of participants
Groups:
- Urea/Lactic Acid Cream: Patients receive topical urea/lactic acid-based cream applied to palms and soles twice daily.
- Placebo Cream: Patients receive placebo cream applied to palms and soles twice daily.
Arm/Group | Urea/Lactic Acid Cream | Placebo Cream
Number analyzed (Participants) | 59 | 49
percentage of participants | 13.6 | 10.2
Statistical Analysis 1: Comparison: Urea/Lactic Acid Cream vs Placebo Cream; Test type: Superiority or Other; p = 0.768, Fisher Exact

2. Secondary Outcome: To Evaluate the Potential Toxicity of Urea/Lactic Acid Cream
Description: Frequency and severity of adverse events reported by patients in weekly diary and evaluated through clinical assessment by NCI CTCAE v3.0. The number of patients reporting grade 3 or higher events are reported in this outcome measure. For a full list of all events, please refer to the Adverse Events section of this report.
Time Frame: Up to 4, 21-day cycles
Population: All patients that were evaluated for adverse events were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Urea/Lactic Acid Cream | Placebo Cream
Number analyzed (Participants) | 67 | 63
participants
  Grade 3+ Adverse Event | 21 | 18
  Grade 4+ Adverse Event | 3 | 3

3. Secondary Outcome: Determine Whether the Prophylactic Use of Vitamin B6 Can Decrease the Incidence and/or Severity of Capecitabine-caused Palmar-plantar Erythrodysesthesia (HFSD).
Description: A patient self-reported hand-foot syndrome diary (HFSD) was completed daily while applying the cream. Patients rated skin severity symptoms individually in their hands and in their feet. Definitions of symptoms, which were based on Common Terminology Criteria for Adverse Events (CTCAE) v3.0, were provided to patients. The number of patients reporting moderate to severe symptoms were tabulated and percentages are reported.
Time Frame: First 3 weeks of treatment
Population: This endpoint is not analyzed due to the fact that Vitamin B6 had already been shown to be ineffective. Additionally, any insignificance may be due to lack of power from the smaller (Arms I, II, III and IV) than target sample size.
Arm/Group | Arm I: (Urea/Lactic Acid +Vit B6) | Arm II: (Urea/Lactic Acid + Placebo) | Arm III: (Placebo +Vit B6) | Arm IV: (Placebo + Placebo) | Arm V: Urea/Lactic Acid | Arm VI: (Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Evaluate the Potential Toxicity of Vitamin B6.
Description: as for outcome 2
Time Frame: up to 4, 21-day cycles
Population: as for outcome 3
Groups:
- Arm IV: (Placebo + Placebo): Patients receive placebo cream as in arm III and oral placebo as in arm II.
Arm/Group | Arm I: (Urea/Lactic Acid +Vit B6) | Arm II: (Urea/Lactic Acid + Placebo) | Arm III: (Placebo +Vit B6) | Arm IV: (Placebo + Placebo) | Arm V: Urea/Lactic Acid | Arm VI: (Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Determine Whether the Prophylactic Use of a Topical Urea/Lactic Acid Cream in Combination With Vitamin B6 Can Decrease the Incidence and/or Severity of Capecitabine Caused Palmar-plantar Erythrodysesthesia.
Description: A patient self-reported hand-foot syndrome diary (HFSD) was completed daily while applying the cream. Patients rated skin severity symptoms individually in their hands and in their feet. Definitions of symptoms, which were based on Common Terminology Criteria for Adverse Events (CTCAE) v3.0, were provided to patients. The number of patients reporting moderate to severe symptoms were tabulated.
Time Frame: First 3 weeks of treatment
Population: as for outcome 3
Groups:
- Arm II: (Urea/Lactic Acid + Placebo): Patients receive topical urea/lactic acid-based cream as in arm I (closed to accrual as of 10/24/2007) and oral placebo once daily on days 1-21.
  urea/lactic acid-based topical cream: Applied topically
  placebo: Given orally or applied topically
- Arm III: (Placebo +Vit B6): Patients receive placebo cream applied to palms and soles twice daily and pyridoxine as in arm I (closed to accrual as of 10/24/2007).
- Arm IV: (Placebo + Placebo): Patients receive placebo cream as in arm III and oral placebo as in arm II (closed to accrual as of 10/24/2007).
Arm/Group | Arm I: (Urea/Lactic Acid +Vit B6) | Arm II: (Urea/Lactic Acid + Placebo) | Arm III: (Placebo +Vit B6) | Arm IV: (Placebo + Placebo) | Arm V: Urea/Lactic Acid | Arm VI: (Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Urea/Lactic Acid Cream | Placebo Cream
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/63
Other Adverse Events (participants affected / at risk) | 56/67 | 50/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urea/Lactic Acid Cream (N=67) | Placebo Cream (N=63)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 26 (39) | 27 (44)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (7) | 5 (6)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Coagulopathy (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 5 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 43 (91) | 34 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less